CLINICAL TRIAL: NCT03455452
Title: A National, Prospective, Non-Interventional Study (NIS) of Nivolumab (BMS-936558) With or Without Ipilimumab (BMS-734016) in Patients With Advanced Renal Cell Carcinoma in Real Life Setting
Brief Title: Non-Interventional Study (NIS) of Nivolumab With or Without Ipilimumab in Participants With Advanced Kidney Cancer
Acronym: WITNESS
Status: Active, not recruiting | Type: Observational
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Other Study IDs: CA209-9GY
Record Dates: First submitted 2018-02-21; First posted 2018-03-06 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Renal Cell Carcinoma; Renal Cell Cancer; Adenocarcinoma Of Kidney; Adenocarcinoma, Renal Cell; Kidney Cancer; Cancer of the Kidney
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Nivolumab: Participants diagnosed with advanced renal cell carcinoma (RCC) and whose physician has decided to initiate a treatment with Nivolumab for the first time for the treatment of RCC
- Cohort 2: Nivolumab + Ipilimumab: Participants diagnosed with advanced RCC and whose physician has decided to start a new systemic therapy with nivolumab + ipilimumab for the first time for the treatment of RCC

SUMMARY:
This is a French, nationwide, prospective, observational, multi-center study in participants diagnosed with advanced renal cell carcinoma, who start a new systemic therapy with nivolumab with or without ipilimumab for the first time and within the market authorization approval.

ELIGIBILITY:
Inclusion Criteria:

-Adult participants with the diagnosis of advanced renal cell cancer (RCC) (histologically or cytologically) whose physician has already decided to initiate a treatment with nivolumab with or without ipilimumab for the first time for the treatment of RCC, according to the label approved in France

NOTE: Nivolumab with ipilimumab is indicated for the first-line treatment of adult participants with intermediate/poor-risk advanced RCC

Exclusion Criteria:

* Primary diagnosis of a cancer other than advanced RCC within the past five years, ie, a cancer other than RCC that requires systemic or other treatment
* Previously treated with anti-PD1, anti-programmed death-ligand 1 (anti-PDL1) or anti-CTLA4 therapy
* Currently included in an interventional clinical trial for advanced or RCC. Participants who have completed participation in an interventional trial; or who are not receiving study drug anymore and who are only followed-up for overall survival (OS) can be enrolled
* Pregnant women and participants under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants who are at least 18 of age at the time of the treatment decision with the diagnosis of advanced renal cell cancer (RCC) (histologically or cytologically confirmed) and whose physician has already decided to initiate a treatment with nivolumab or with nivolumab plus ipilimumab for the first time for the treatment of RCC, according to the label approved in France.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2018-01-21 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 3 years
  By Cohort

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 3 years
Progression Free Survival (PFS) | Up to 3 years
Overall Response Rate (ORR) | Up to 3 years
Best Overall Response Rate (BORR) | Up to 3 years
Best Overall Response (BOR) | Up to 3 years
Distribution of socio-demographic characteristics of participants | Approximately 3 years
Distribution of clinical characteristics of participants | Approximately 3 years
Distribution of management of participants with treatment-related adverse events (AEs) | Approximately 3 years
Distribution of management of participants according to Memorial Sloan Kettering Cancer Center (MSKCC) score | At baseline
Distribution of management of participants according to International Metastatic Renal Cell Carcinoma Database Consortium (IMDC) score | At baseline
Distribution of treatment patterns in participants with advanced Renal Cell Carcinoma (RCC) | Approximately 3 years
Distribution of incidence of AEs | Approximately 3 years
Distribution of Severity of AEs | Approximately 3 years
Distribution of management of AEs | Approximately 3 years
Health-related quality of life of participants using Functional Assessment of Cancer Therapy -Kidney Symptom Index (FKSI-19) questionnaires | Approximately 3 years
  The FKSI-19 will be graded by the patient on a scale from 0 to 4 (range "not at all to very much")
Health-related quality of life of participants using European Quality of Life-5 Dimensions (EQ-5D) questionnaires | Approximately 3 years
  The EQ-5D descriptive system consists of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression, each with 3 levels (eg, no problems, moderate problems, extreme problems)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Paris, France

REFERENCES:
- [Derived] Barthelemy P, Albiges L, Escudier B, Narciso B, Bigot P, Chehimi M, Emambux S, Calcagno F, Mouillet G, Eymard JC, Schlurmann F, Bailly S, Garbay D, Berdah JF, Palmaro MB, Goupil MG, Spaeth D, Nere S, Quentric C, Vano YA, Thiery-Vuillemin A. Nivolumab in patients with advanced renal cell carcinoma in France: interim results of the observational, real-world WITNESS study. ESMO Open. 2024 Jul;9(7):103602. doi: 10.1016/j.esmoop.2024.103602. Epub 2024 Jun 18. PMID 38897136
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html